CLINICAL TRIAL: NCT01051180
Title: Haemorrhoidal Artery Ligation Operation; is Doppler Necessary?
Brief Title: Is Doppler Necessary in Haemorrhoidal Artery Ligation Operation?
Status: Terminated | Type: Observational
Why Stopped: Doppler device company wanted hospital to stop recruiting
Sponsor: Poole Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Guy Nash, Consultant Surgeon, Poole Hospital NHS Foundation Trust
Other Study IDs: 09/H0501/61
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Piles; Bleeding
Keywords: HEMORRHOIDS; TREATMENT; PILES; BLEEDING; HALO
MeSH Terms: conditions — Hemorrhoids; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Doppler: Those patients where the doppler was randomised to be on
  Interventions: Procedure: HALO
- Non doppler patients: those with no doppler guidance
  Interventions: Procedure: HALO

INTERVENTIONS:
Procedure: HALO — Ligation of haemorrhoidal arteries

SUMMARY:
Haemorrhoidal artery ligation operation (HALO) is an operation that ties off vessels to piles. This study examines whether the ultrasound (doppler) is necessary to guide this tying off or not.

DETAILED DESCRIPTION:
HALO (haemorrhoidal artery ligation operation) has proved to be a popular and effective treatment for bleeding piles. Currently the HALO is a Doppler guided procedure though when the Doppler mechanism does not function it has been noted that the results are similar. This prompts the question does the Doppler guide the operation to tie off the important vessels to shrink he piles, or can the vessels that underlie the visible piles be treated without Doppler. Professor Phillips from St.Marks has reviewed the protocol and agrees that it is well designed and worthwhile.

ELIGIBILITY:
Inclusion Criteria:

* For consenting adults (18-90 years) with grade one and two piles listed for HALO at Poole hospital by three consultants trained in the HALO technique, the patients will be offered to be involved in the study.

Exclusion Criteria:

* Other grades of piles, age outside 18-90 or other anal condition

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For consenting adults (18-90 years) with grade one and two piles listed for HALO at Poole hospital by three consultants trained in the HALO technique, the patients will be offered to be involved in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Improvement of rectal bleeding | 3-6 months

SECONDARY OUTCOMES:
Satisfaction with the HALO procedure with or without doppler guidance | 3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Poole Hospital, Poole, Dorset, United Kingdom